CLINICAL TRIAL: NCT05221515
Title: The Effectiveness of an Attention-based Intervention for School Aged Autistic Children With Anger Regulating Problems: a Randomized Controlled Trial
Brief Title: The Effectiveness of an Attention-based Intervention for School Aged Autistic Children With Anger Regulating Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Sander Begeer, Professor, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOBpaper2021
Record Dates: First submitted 2021-11-23; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; Anger; Randomized controlled trial
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention condition (Experimental): Participants received both parent training and child-focussed treatment
  Interventions: Behavioral: Anger can go!; Behavioral: Parent psycho-education
- Control condition (Active Comparator): Participants received only parent training
  Interventions: Behavioral: Parent psycho-education

INTERVENTIONS:
Behavioral: Anger can go! — The intervention "Anger Can Go!" was designed to treat anger regulation problems in autistic children aged 8 to 13 years old. The intervention consists of nine sessions of 60 minutes and is divided in four phases. Phase 1: psycho-education, affect-education and measuring anger with an anger-thermometer. This is a self-report scale presented as the drawing of a thermometer, that allows the child to indicate his level of anger, as linked to specific bodily and behavioral representations on a scale from 0 to 3. Phase 2: making a functional behavior assessment (FBA) and taking a time-out at a low anger-level (between 1 and 2 on the scale 0 to 3) to prevent aggressive outbursts. Phase 3: taking a time-out at a low anger-level (between 1 and 2 on the scale 0 to 3) to prevent aggressive outbursts, shifting attention away from aversive stimuli, to cope with the stress of the anger provoking situation. Phase 4: creating solutions to cope with an anger provoking situation.
  Arms: Intervention condition
Behavioral: Parent psycho-education — Three psycho-educational parent group sessions (take place before the children's sessions in intervention group). Parents meet with other parents and a therapist to learn about the nature of their Expressed Emotion (EE) and how it relates to the child's aggressive behavior.

SUMMARY:
Children on the autism spectrum often show aggressive behavior. Treatment can train children to be more aware of their emotions. Investigators studied the effectiveness of an attention-based intervention tailored on aggressive behavior problems and the use of anger coping strategies of school aged autistic children with anger regulation problems.

DETAILED DESCRIPTION:
Investigators studied the effectiveness of an attention-based intervention tailored on aggressive behavior problems and the use of anger coping strategies of school aged autistic children with anger regulation problems. Using a randomized controlled trial (RCT), children were allocated to the attention-based treatment in combination with a psycho-educational parent-training (treatment group) or to the parent-training only (active control group).

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of autism spectrum disorder
* age 8 - 13
* seeking treatment for aggressive behaviour problems

Exclusion Criteria:

* psychotropic medication still being set

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Aggressive behavior problems: Arguing, Temper tantrums, Destroying things and Physical violence | At week 0, before the intervention group received treatment
  Questionnaire Social Behavior (QSB) measuring behavioral and emotion regulation problems typical for autistic children.
Aggressive behavior problems: Arguing, Temper tantrums, Destroying things and Physical violence | 9 weeks later after treatment
  Questionnaire Social Behavior (QSB) measuring behavioral and emotion regulation problems typical for autistic children.
Aggressive behavior problems: aggression as reported by parent | At week 0, before the intervention group received treatment
  The aggression sub scale from the Child Behavior Checklist (CBCL). Minimum value: 0, maximum value: 36. A higher score means more aggression.
Aggressive behavior problems: aggression as reported by parent | 9 weeks later after treatment
  The aggression sub scale from the Child Behavior Checklist (CBCL). Minimum value: 0, maximum value: 36. A higher score means more aggression.
Aggressive behavior problems: aggression as reported by teacher | At week 0, before the intervention group received treatment
  The aggression sub scale from the Teacher Rating Form (TRF). Minimum value: 0, maximum value: 36. A higher score means more aggression.
Aggressive behavior problems: aggression as reported by teacher | 9 weeks later after treatment
  The aggression sub scale from the Teacher Rating Form (TRF). Minimum value: 0, maximum value: 36. A higher score means more aggression.
Anger coping strategies | At week 0, before the intervention group received treatment
  The Behavioral Anger Response Questionnaire for children (BARQ-C)
Anger coping strategies | 9 weeks later after treatment
  The Behavioral Anger Response Questionnaire for children (BARQ-C)

SECONDARY OUTCOMES:
Quality of life of the child | At week 0, before the intervention group received treatment
  Pediatric Quality of life inventory (Peds ql): Physical Functioning, Emotional Functioning, Social Functioning and School Functioning.
Quality of life of the child | 9 weeks later after treatment
  Pediatric Quality of life inventory (Peds ql): Physical Functioning, Emotional Functioning, Social Functioning and School Functioning.
Social impairment due to autism symptoms | At week 0, before the intervention group received treatment
  Social Responsiveness Scale (SRS). Minimum value: 0, maximum value: 195. A higher score means more impairments.
Social impairment due to autism symptoms | 9 weeks later after treatment
  Social Responsiveness Scale (SRS). Minimum value: 0, maximum value: 195. A higher score means more impairments.
Parental stress | At week 0, before the intervention group received treatment
  Nijmeegse Ouderlijke Stress Index (NOSI). Minimum value: 6, maximum value: 66. A higher score means more stress
Parental stress | 9 weeks later after treatment
  Nijmeegse Ouderlijke Stress Index (NOSI). Minimum value: 6, maximum value: 66. A higher score means more stress
Parental well-being | At week 0, before the intervention group received treatment
  Symptom Checklist-90 (SCL-90). Minimum value: 0, maximum value: 360. A higher score indicates a worse well-being.
Parental well-being | 9 weeks later after treatment
  Symptom Checklist-90 (SCL-90). Minimum value: 0, maximum value: 360. A higher score indicates a worse well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Frits Boer, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - De Bascule, Amsterdam, North Holland
  - Wei43, Amsterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carr, E. G., & Horner, R. H. (2007). The expanding vision of positive behavior support: Research perspectives on happiness, helpfulness, hopefulness. Journal of positive behavior interventions, 9(1), 3-14.
- [Background] Chalfant AM, Rapee R, Carroll L. Treating anxiety disorders in children with high functioning autism spectrum disorders: a controlled trial. J Autism Dev Disord. 2007 Nov;37(10):1842-57. doi: 10.1007/s10803-006-0318-4. Epub 2006 Dec 15. PMID 17171539
- [Background] Fung LK, Mahajan R, Nozzolillo A, Bernal P, Krasner A, Jo B, Coury D, Whitaker A, Veenstra-Vanderweele J, Hardan AY. Pharmacologic Treatment of Severe Irritability and Problem Behaviors in Autism: A Systematic Review and Meta-analysis. Pediatrics. 2016 Feb;137 Suppl 2:S124-35. doi: 10.1542/peds.2015-2851K. PMID 26908468
- [Background] Goel R, Hong JS, Findling RL, Ji NY. An update on pharmacotherapy of autism spectrum disorder in children and adolescents. Int Rev Psychiatry. 2018 Feb;30(1):78-95. doi: 10.1080/09540261.2018.1458706. Epub 2018 Apr 25. PMID 29693461
- [Background] Gross, J. J. (2015). Emotion regulation: Current status and future prospects. Psychological inquiry, 26(1), 1-26.
- [Background] Hartmann K, Urbano MR, Raffaele CT, Kreiser NL, Williams TV, Qualls LR, Elkins DE. Outcomes of an emotion regulation intervention group in young adults with autism spectrum disorder. Bull Menninger Clin. 2019 Summer;83(3):259-277. doi: 10.1521/bumc.2019.83.3.259. PMID 31502871
- [Background] Ibrahim K, Kalvin C, Marsh CL, Anzano A, Gorynova L, Cimino K, Sukhodolsky DG. Anger Rumination is Associated with Restricted and Repetitive Behaviors in Children with Autism Spectrum Disorder. J Autism Dev Disord. 2019 Sep;49(9):3656-3668. doi: 10.1007/s10803-019-04085-y. PMID 31144231
- [Background] Kanne SM, Mazurek MO. Aggression in children and adolescents with ASD: prevalence and risk factors. J Autism Dev Disord. 2011 Jul;41(7):926-37. doi: 10.1007/s10803-010-1118-4. PMID 20960041
- [Background] Linehan, M. (2014). DBT? Skills training manual. Guilford Publications.
- [Background] Luiselli, J. K. (Ed.). (2014). Children and youth with autism spectrum disorder (ASD): recent advances and innovations in assessment, education, and intervention.
- [Background] Mascha, K., & Boucher, J. (2006). Preliminary investigation of a qualitative method of examining siblings' experiences of living with a child with ASD. The British Journal of Development Disabilities, 52(102), 19-28.
- [Background] McStay RL, Dissanayake C, Scheeren A, Koot HM, Begeer S. Parenting stress and autism: the role of age, autism severity, quality of life and problem behaviour of children and adolescents with autism. Autism. 2014 Jul;18(5):502-10. doi: 10.1177/1362361313485163. Epub 2013 Oct 8. PMID 24104515
- [Background] Mazurek, M. O., Kanne, S. M., & Wodka, E. L. (2013). Physical aggression in children and adolescents with autism spectrum disorders. Research in Autism Spectrum Disorders, 7(3), 455-465.
- [Background] Patel S, Day TN, Jones N, Mazefsky CA. Association between anger rumination and autism symptom severity, depression symptoms, aggression, and general dysregulation in adolescents with autism spectrum disorder. Autism. 2017 Feb;21(2):181-189. doi: 10.1177/1362361316633566. Epub 2016 Jul 9. PMID 27095831
- [Background] Hill AP, Zuckerman KE, Hagen AD, Kriz DJ, Duvall SW, van Santen J, Nigg J, Fair D, Fombonne E. Aggressive Behavior Problems in Children with Autism Spectrum Disorders: Prevalence and Correlates in a Large Clinical Sample. Res Autism Spectr Disord. 2014 Sep 1;8(9):1121-1133. doi: 10.1016/j.rasd.2014.05.006. PMID 25221619
- [Background] Reese RM, Richman DM, Belmont JM, Morse P. Functional characteristics of disruptive behavior in developmentally disabled children with and without autism. J Autism Dev Disord. 2005 Aug;35(4):419-28. doi: 10.1007/s10803-005-5032-0. PMID 16134028
- [Background] Samson AC, Phillips JM, Parker KJ, Shah S, Gross JJ, Hardan AY. Emotion dysregulation and the core features of autism spectrum disorder. J Autism Dev Disord. 2014 Jul;44(7):1766-72. doi: 10.1007/s10803-013-2022-5. PMID 24362795
- [Background] Samson AC, Wells WM, Phillips JM, Hardan AY, Gross JJ. Emotion regulation in autism spectrum disorder: evidence from parent interviews and children's daily diaries. J Child Psychol Psychiatry. 2015 Aug;56(8):903-13. doi: 10.1111/jcpp.12370. Epub 2014 Dec 1. PMID 25442191
- [Background] Segal, Z. V., Williams, J. M. G., & Teasdale, J. D. (2013). Mindfulness-based cognitive therapy for depression. Guilford Publications.
- [Background] Sofronoff K, Attwood T, Hinton S, Levin I. A randomized controlled trial of a cognitive behavioural intervention for anger management in children diagnosed with Asperger syndrome. J Autism Dev Disord. 2007 Aug;37(7):1203-14. doi: 10.1007/s10803-006-0262-3. PMID 17082978
- [Background] Wong C, Odom SL, Hume KA, Cox AW, Fettig A, Kucharczyk S, Brock ME, Plavnick JB, Fleury VP, Schultz TR. Evidence-Based Practices for Children, Youth, and Young Adults with Autism Spectrum Disorder: A Comprehensive Review. J Autism Dev Disord. 2015 Jul;45(7):1951-66. doi: 10.1007/s10803-014-2351-z. PMID 25578338
- [Background] White SW, Ollendick T, Scahill L, Oswald D, Albano AM. Preliminary efficacy of a cognitive-behavioral treatment program for anxious youth with autism spectrum disorders. J Autism Dev Disord. 2009 Dec;39(12):1652-62. doi: 10.1007/s10803-009-0801-9. Epub 2009 Jun 30. PMID 19568924
- [Background] White SW, Albano AM, Johnson CR, Kasari C, Ollendick T, Klin A, Oswald D, Scahill L. Development of a cognitive-behavioral intervention program to treat anxiety and social deficits in teens with high-functioning autism. Clin Child Fam Psychol Rev. 2010 Mar;13(1):77-90. doi: 10.1007/s10567-009-0062-3. PMID 20091348
- [Background] Wood JJ, Drahota A, Sze K, Har K, Chiu A, Langer DA. Cognitive behavioral therapy for anxiety in children with autism spectrum disorders: a randomized, controlled trial. J Child Psychol Psychiatry. 2009 Mar;50(3):224-34. doi: 10.1111/j.1469-7610.2008.01948.x. PMID 19309326
- [Result] Bos MGN, Diamantopoulou S, Stockmann L, Begeer S, Rieffe C. Emotion Control Predicts Internalizing and Externalizing Behavior Problems in Boys With and Without an Autism Spectrum Disorder. J Autism Dev Disord. 2018 Aug;48(8):2727-2739. doi: 10.1007/s10803-018-3519-8. PMID 29512017
- [Result] Dempsey AG, Llorens A, Brewton C, Mulchandani S, Goin-Kochel RP. Emotional and behavioral adjustment in typically developing siblings of children with autism spectrum disorders. J Autism Dev Disord. 2012 Jul;42(7):1393-402. doi: 10.1007/s10803-011-1368-9. PMID 21984214
- [Result] Fernandez-Alcantara M, Garcia-Caro MP, Perez-Marfil MN, Hueso-Montoro C, Laynez-Rubio C, Cruz-Quintana F. Feelings of loss and grief in parents of children diagnosed with autism spectrum disorder (ASD). Res Dev Disabil. 2016 Aug;55:312-21. doi: 10.1016/j.ridd.2016.05.007. Epub 2016 May 25. PMID 27235768
- [Result] Mazefsky CA, Kao J, Oswald DP. Preliminary evidence suggesting caution in the use of psychiatric self-report measures with adolescents with high-functioning autism spectrum disorders. Res Autism Spectr Disord. 2011 Jan;5(1):164-174. doi: 10.1016/j.rasd.2010.03.006. PMID 24013401
- [Result] Ridderinkhof A, de Bruin EI, Blom R, Bogels SM. Mindfulness-Based Program for Children with Autism Spectrum Disorder and Their Parents: Direct and Long-Term Improvements. Mindfulness (N Y). 2018;9(3):773-791. doi: 10.1007/s12671-017-0815-x. Epub 2017 Oct 6. PMID 29875881
- [Result] Singh, N. N., Lancioni, G. E., Manikam, R., Winton, A. S., Singh, A. N., Singh, J., & Singh, A. D. (2011). A mindfulness-based strategy for self-management of aggressive behavior in adolescents with autism. Research in Autism Spectrum Disorders, 5(3), 1153-1158.
- [Result] Seymour M, Wood C, Giallo R, Jellett R. Fatigue, stress and coping in mothers of children with an autism spectrum disorder. J Autism Dev Disord. 2013 Jul;43(7):1547-54. doi: 10.1007/s10803-012-1701-y. PMID 23124359
- [Result] Shivers CM, Jackson JB, McGregor CM. Functioning Among Typically Developing Siblings of Individuals with Autism Spectrum Disorder: A Meta-Analysis. Clin Child Fam Psychol Rev. 2019 Jun;22(2):172-196. doi: 10.1007/s10567-018-0269-2. PMID 30178117
- [Result] Spek AA, van Ham NC, Nyklicek I. Mindfulness-based therapy in adults with an autism spectrum disorder: a randomized controlled trial. Res Dev Disabil. 2013 Jan;34(1):246-53. doi: 10.1016/j.ridd.2012.08.009. Epub 2012 Sep 8. PMID 22964266
- [Result] Tanksale R, Sofronoff K, Sheffield J, Gilmour J. Evaluating the effects of a yoga-based program integrated with third-wave cognitive behavioral therapy components on self-regulation in children on the autism spectrum: A pilot randomized controlled trial. Autism. 2021 May;25(4):995-1008. doi: 10.1177/1362361320974841. Epub 2020 Nov 25. PMID 33238718
- [Result] Zaidman-Zait A, Mirenda P, Duku E, Vaillancourt T, Smith IM, Szatmari P, Bryson S, Fombonne E, Volden J, Waddell C, Zwaigenbaum L, Georgiades S, Bennett T, Elsabaggh M, Thompson A. Impact of personal and social resources on parenting stress in mothers of children with autism spectrum disorder. Autism. 2017 Feb;21(2):155-166. doi: 10.1177/1362361316633033. Epub 2016 Jul 9. PMID 27091948